CLINICAL TRIAL: NCT00474669
Title: A Phase I Study of Intraperitoneal Hyperthermic Docetaxel at the Time of Second Look Surgery Following Front-Line Normothermic Intraperitoneal and Intravenous Cisplatin/Paclitaxel for Patients With Stage II and III Ovarian Carcinoma
Brief Title: A Phase I Study of Intraperitoneal Hyperthermic Docetaxel
Acronym: IP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCC-GYN-07-001
Record Dates: First submitted 2007-05-15; First posted 2007-05-17 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Ovarian Carcinoma
Keywords: Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel (Experimental): Intraperitoneal Docetaxel administered with heat
  Interventions: Drug: docetaxel

INTERVENTIONS:
Drug: docetaxel — Docetaxel will be administered in normal-saline delivered at an inflow temperature of 42 degreesC for 90 minutes by the technique described in Appendix D of the protocol

SUMMARY:
The primary objective is to assess the maximum tolerated dose of docetaxel administered intraperitoneally with heat at the time of second-look surgery in patients with stage II/III ovarian carcinoma.

DETAILED DESCRIPTION:
This is a phase I study of intraperitoneal hyperthermic docetaxel given at the time of second look surgery following front-line normothermic intraperitoneal and intravenous cisplatin/paclitaxel for patients with stage II and III ovarian carcinoma. The primary objectives are to assess the maximum tolerated dose of docetaxel administered intraperitoneally with heat at this time and assess the toxicity and morbidity associated with this treatment. Eligible patients will have had a complete clinical response to front-line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had a complete clinical response (negative clinical examination, CA125 and CT scan of chest, abdomen and pelvis) to front-line therapy for stage II/III ovarian, primary peritoneal or Fallopian tube carcinoma. This will have included initial surgery followed by combined IV/IP chemotherapy with cisplatin and paclitaxel. Patients must have had a minimum of three courses of IP therapy with both paclitaxel and cisplatin
* Second surgery to be performed no more than 3 months from last course of initial chemotherapy
* Age greater than 18 years and negative pregnancy if has child-bearing potential
* GOG performance status less than 2
* Medically fit for surgery
* Patients must have normal organ and marrow function as defined in the protocol hepatic function Total Bilirubin ULN AST and ALT and Alkaline Phosphatase must be within the range allowing for eligibility. In determining eligibility the more abnormal of the two values AST or ALT) should be used.
* Ability to understand and the willingness to sign a written informed consent document.
* The effects of docetaxel on the developing human fetus are unknown. For this reason and because taxanes are known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

* Patients who have completed front-line therapy for ovarian cancer more than 3 months prior to HIPEC.
* Patients receiving any other investigational agents.
* Patients with stage IV disease including previous parenchymal liver disease, brain metastasis or cytologically-confirmed chest metastasis
* Patients with a history of severe hypersensitivity reaction to Taxotere® or other drugs formulated with polysorbate 80. History of allergic reactions attributed to compounds of similar chemical or biologic composition used in this study in addition to Taxotere.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* More than grade 2 peripheral neuropathy from prior chemotherapy
* Pregnant, breast-feeding or known to be HIV positive
* Prior malignancy other than non-melanomatous skin cancer more than 5 years ago
* No prior chemotherapy other than for front-line ovarian cancer or radiation for any reason.
* Stomatitis of any grade
* Uncontrolled intercurrent illness or other conditions that would limit compliance with study requirements should be excluded.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Assess the MTD of docetaxel administered intraperitoneally with heat at the time of second-look surgery in patients with stage II/III ovarian carcinoma following surgery and normothermic intraperitoneal and intravenous cisplatin and paclitaxel. | 6 months-5 years

SECONDARY OUTCOMES:
To assess the quality of life of patients treated with intraperitoneal hyperthermic chemotherapy in this setting | 6 months-5 years

CONTACTS AND LOCATIONS:
Overall Officials: C. William Helm, MD, Principal Investigator — James Graham Brown Cancer Center
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States

REFERENCES:
- [Result] 1 - R. Bruno, D. Hille, L. Thomas, A. Riva and L.B. Sheiner. Population Pharmacokinetics / Pharmacodynamics (PK/PD) of Docetaxel (Taxotere) in Phase II studies. Proc. ASCO, 14, 457, 1995. 2 - S. L. Beal, A.J. Boeckman and L.B. Sheiner. NONMEM version 4. User's Guide Part I to VI. University of California at San Francisco, San Francisco, 1988 - 1992.